CLINICAL TRIAL: NCT03522285
Title: Outcome of Total Hip Replacement in Patients With Chronic Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MBMady, resident of orthopedics and trauma surgery, Assiut University
Other Study IDs: hip arthroplasty
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Arthroplasty Complications
Keywords: hip arthroplasty; chronic renal diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: investigation: erythrocyte sedimentation rate — investigations will be done to detect presence of infection and x-ray also for detection of infection or loosing of hip components
  Other Names: radiation: x-ray; investigation: C reactive protein; investigation: complete blood count

SUMMARY:
the study aims to determine rate of mortality and morbidity after total hip replacement in patients with chronic kidney diseases and incidence of periprosthetic joint infection in these patients.

DETAILED DESCRIPTION:
Retrospective review of the database of arthroplasty unit was conducted from January 2014 to December 2018. Data of all patients who suffered from chronic kidney disease and underwent hip arthroplasty because of fracture neck of femur or arthritis or head necrosis or any other cause , will be collected as, Demographic characteristics: age , gender , place of residence and diagnosis. Medical comorbidities: other comorbidities will be taken in consideration as Diabetes, Hypertension and cardiac problems.

Detailed history of patient's renal disease: cause of renal disease ,duration of the renal disease , grading of renal failure according to National Kidney Foundation (NKF) guidelines , medical treatment : whether the patient is on regular medical treatment or not, duration of medical treatment and type of medications and dialysis history : whether the patient is dialysis dependant or not, duration of being dialysis dependant and frequency of dialysis.

Post operative surgical complications as : dislocation, infection , periprosthetic fracture or loosing and osteolysis.

Post operative medical complications as : myocardial infarction , stroke , pulmonary embolism and deep venous thrombosis.

At Follow up :

Clinical assessment will be done for signs of infection as hotness , redness, tenderness and discharge from wound site.

Functional assessment also will be done , it will be done by Harris Hip Score (HHS), Hip Disability and Osteoarthritis Outcome Score (HOOS) and The 12-Item Short Form Survey (SF-12).

Radiological assessment also will be done for signs of loosing as lucency and component migration and for signs of infection as periosteal reaction , irregular osteolysis , absence of sclerotic border and cortical bone resorption .

Investigations for periprosthetic infection will be carried out: erythrocyte sedimentation rate (ESR), C- reactive protein (CRP) and complete blood count (CBC) to predict presence of infection , if they are positive , aspiration will be carried out to know type of organism.

If there is past definite history of infection, detailed data will be recorded as:

Time of presence of infection from surgery and result of culture and sensitivity ( if was done) to know the type of the organism,type of treatment done(whatever medical or surgical treatment) and frequency of infection recurrence.

Also history of revision surgery , rate and its causes will be recorded.

Those patients will be divided into two groups, one group is that group of chronic renal disease patients who were on regular dialysis at time of operation and the other is that group who were not dialysis dependant at time of operation . rate of each complication of the previously mentioned complications, will be calculated in the two groups . Results will show which group is at higher risk of complications of the two groups .

ELIGIBILITY:
Inclusion Criteria:

1. patients with chronic renal disease who had total hip arthroplasty .
2. Patients underwent hip arthroplasty between January 2014 to December 2017 in Assiut University Hospital

Exclusion Criteria:

No patients will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic renal diseases who underwent total hip replacement surgery from January 2014 to December 2017
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity and mortality after total hip replacement in patients with chronic kidney disease | one year

SECONDARY OUTCOMES:
Incidence of periprosthetic infection after total hip replacement in patients with chronic renal diseases; dialysis dependant and non- dependant | one year
  rate of incidence of periprosthetic infection after total hip replacement in patients with chronic renal diseases, frequency of recurrence of infection and if dialysis dependency increase risk of infection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levey AS, Beto JA, Coronado BE, Eknoyan G, Foley RN, Kasiske BL, Klag MJ, Mailloux LU, Manske CL, Meyer KB, Parfrey PS, Pfeffer MA, Wenger NK, Wilson PW, Wright JT Jr. Controlling the epidemic of cardiovascular disease in chronic renal disease: what do we know? What do we need to learn? Where do we go from here? National Kidney Foundation Task Force on Cardiovascular Disease. Am J Kidney Dis. 1998 Nov;32(5):853-906. doi: 10.1016/s0272-6386(98)70145-3. No abstract available. PMID 9820460
- [Background] Ayers DC, Athanasou NA, Woods CG, Duthie RB. Dialysis arthropathy of the hip. Clin Orthop Relat Res. 1993 May;(290):216-24. PMID 8472452
- [Background] Tejwani NC, Schachter AK, Immerman I, Achan P. Renal osteodystrophy. J Am Acad Orthop Surg. 2006 May;14(5):303-11. doi: 10.5435/00124635-200605000-00006. PMID 16675624
- [Background] DiRaimondo CR, Casey TT, DiRaimondo CV, Stone WJ. Pathologic fractures associated with idiopathic amyloidosis of bone in chronic hemodialysis patients. Nephron. 1986;43(1):22-7. doi: 10.1159/000183712. PMID 3703063
- [Background] Gualtieri G, Vellani G, Dallari D, Catamo L, Gualtieri I, Fatone F, Bonomini V. Total hip arthroplasty in patients dialyzed or with renal transplants. Chir Organi Mov. 1995 Apr-Jun;80(2):139-45. English, Italian. PMID 7587515
- [Background] McCleery MA, Leach WJ, Norwood T. Rates of infection and revision in patients with renal disease undergoing total knee replacement in Scotland. J Bone Joint Surg Br. 2010 Nov;92(11):1535-9. doi: 10.1302/0301-620X.92B11.23870. PMID 21037348
- [Background] Deo S, Gibbons CL, Emerton M, Simpson AH. Total hip replacement in renal transplant patients. J Bone Joint Surg Br. 1995 Mar;77(2):299-302. PMID 7706352
- [Background] Bradford DS, Janes PC, Simmons RS, Najarian JS. Total hip arthroplasty in renal transplant recipients. Clin Orthop Relat Res. 1983 Dec;(181):107-14. PMID 6357584